CLINICAL TRIAL: NCT00251238
Title: Efficacy and Tolerability of Ginkgo Biloba Extract EGb 761® in Patients With Raynaud´s Phenomenon
Brief Title: Efficacy and Tolerability of Ginkgo Biloba Extract in Patients With Raynaud´s Phenomenon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VSM Geneesmiddelen b.v. (Industry)
Responsible Party: Principal Investigator, Sebastian JH Bredie, MD, PhD, SJH Bredie, internist, MD, PhD, VSM Geneesmiddelen b.v.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 523052.01.002
Record Dates: First submitted 2005-11-08; First posted 2005-11-09 (Estimated); Results first posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Raynaud Disease
Keywords: Raynaud´s phenomenon; Vasospastic attacks; Ginkgo biloba
MeSH Terms: conditions — Raynaud Disease | interventions — Ginkgo biloba extract; Ginkgo Extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ginkgo biloba extract EGb 761 (Experimental): Receiving daily Ginkgo biloba extract EGb 761
  Interventions: Drug: Ginkgo biloba extract EGb 761
- Placebo (Placebo Comparator): Receiving daily placebo
  Interventions: Drug: Ginkgo biloba extract EGb 761

INTERVENTIONS:
Drug: Ginkgo biloba extract EGb 761 — daily Ginkgo biloba extract EGb 761
  Other Names: Ginkgo biloba

SUMMARY:
The aim of the study is to investigate the efficacy and safety of EGb 761® in patients with the primary Raynaud phenomenon, with regards to the frequency, duration and severity of vasospastic attacks.

DETAILED DESCRIPTION:
Despite more than 150 years of research into the pathophysiology of Raynaud´s phenomenon it is still not understood sufficiently. Three mean mechanisms responsible for Raynaud´s phenomenon are discussed and fall into the following three categories:

* neurological malfunction
* pathological blood vessel wall and blood cell interactions
* inflammatory and immunological responses Based on these concepts different classes of drugs have been tested. Although some therapies have shown effects, prolongation of the therapy is often difficult due to side-effects.

Considering a prevalence of 5-10% in the general population, there is still a place and probably a need for the development of new treatment concepts. Ginkgo biloba has shown to have anti-oxidative and anti-platelet activities. In a small placebo controlled trial in patients with the Raynaud´s phenomenon promising results for the Ginkgo biloba extract were shown. EGb 761® is known to be safe and well tolerated. Based on the above considerations, EGb 761® may be an effective treatment for Raynaud´s phenomenon.

Aim: To determine the efficacy and safety of EGb 761® in patients with Raynaud´s phenomenon on the frequency, duration, and severity of vasospastic attacks compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Primary Raynaud´s phenomenon
* History of episodic digital or toe pallor
* Duration of Raynaud´s phenomenon at least 2 years
* Suffering form regular occuring attacks prior to enrolment

Exclusion Criteria:

* Secondary Raynaud´s phenomenon
* Connective tissue disease
* Large vessel disease
* Cryoglobulinemia, cold agglutinins disease, thrombocytosis
* Concomitant pharmacological treatment with effects on the vasculature
* Pregnancy or lactation
* Severe internal or systemic disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-11; Primary Completion 2006-03 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Department, Study Director — VSM Geneesmiddelen b.v.
Locations (1):
- UMC ST Radboud, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: active treatment group, receiving oral film-coated tablet of 120-mg Ginkgo Biloba special extract (EGb 761) 2 times a day for 10 weeks, after an initial 2-week run-in phase
- Placebo Group: receiving matching placebo
Period: Overall Study
Arm/Group | Intervention Group | Placebo Group
Started | 21 | 20
Completed | 21 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: active treatment group, receiving film coated 120 mg Ginkgo Biloba special extract (EGb 761) two times a day for 10 weeks
- Control Group: Receiving matching placebo
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 39
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (13) | 49 (13) | 48 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  Netherlands | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Vasospastic Attacks
Time Frame: Number of Vasospastic Attacks per day, for up to 10 weeks
Measure: Mean (Standard Deviation); unit: attacks per day
Groups:
- Intervention Group: active treatment group (EGb 761)
- Placebo Group: receiving placebo
Arm/Group | Intervention Group | Placebo Group
Number analyzed (Participants) | 21 | 20
attacks per day | 2.4 (2.6) | 2.0 (1.8)

2. Primary Outcome: Duration of Vasospastic Attacks
Time Frame: minutes per day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention Group | Placebo Group
Number analyzed (Participants) | 21 | 20
minutes | 47.4 (63.0) | 50.9 (84.7)

3. Primary Outcome: Change From Baseline in Severity of Vasospastic Attacks
Description: Severity of the complains due to Vasospastic Attacks was measured using a 10-steps likert scale.
  The scale ranged between 0 and 10, with higher scores indicating more severe attacks.
Time Frame: Baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Placebo Group
Number analyzed (Participants) | 21 | 20
units on a scale | -1.3 (2.3) | -1.3 (2.4)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 3/21 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=21) | Placebo Group (N=20)
headache (Nervous system disorders) | 2 (2) | 2 (2)
dyspnoe (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No